CLINICAL TRIAL: NCT04365517
Title: The Effect of Sitagliptin Treatment in COVID-19 Positive Diabetic Patients
Acronym: SIDIACO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Director of Endocrinology and Diabetology ASST FBF Sacco, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sacco FBF
Record Dates: First submitted 2020-04-14; First posted 2020-04-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Diabetes Mellitus, Type 2; CKD
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: A randomized controlled open label intervention study is proposed. Patients hospitalized for COVID-19 and suffering from type 2 diabetes will be included in the study and divided into two groups by randomization: sitagliptin add-on therapy with nutritional therapy with or without insulin (study group) vs nutritional therapy with or without insulin (group of control, standard therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Active Comparator): patients will be treated with sitagliptin add on to nutritional therapy with o without insulin treatment. The dose of sitagliptin will be established on the basis of the estimated glomerular filtrate: 100 mg in single daily administration (estimated glomerular filtration rate less than or equal to 45 mL / min / 1.73 m2) or 50 mg (estimated glomerular filtration rate 30-45 mL / min / 1.73 m2) in combination or not with insulin. Patients with stage IV and V renal failure (estimated glomerular filtration rate less than or equal to 30 mL / min / 1.73 m2) will be excluded
  Interventions: Drug: Sitagliptin
- Control group (No Intervention): Patients who will be prescribed nutritional therapy with or without insulin treatment

INTERVENTIONS:
Drug: Sitagliptin — We propose a randomized controlled open label intervention study. Patients with type 2 diabetes admitted to COVID-19 and randomized to the study group will be treated with sitagliptin at an adjusted dosage for estimated glomerular filtrate: 100 mg once daily (estimated glomerular filtration rate less than or equal to 45 mL / min / 1.73 m2 ) or 50 mg (estimated glomerular filtration rate 30-45 mL / min / 1.73 m2) in combination or not with insulin. Patients with stage IV and V renal failure (estimated glomerular filtration rate less than or equal to 30 mL / min / 1.73 m2) will be excluded
  Arms: Treatment group

SUMMARY:
The COVID-19 pathology is frequently associated with diabetes mellitus and metabolic syndrome. In the epidemic outbreak that exploded at the beginning of 2020 in the Lombardy Region, about two thirds of the patients who died from COVID-19 were affected by diabetes mellitus. COVID-19 occurs in 70% of cases with an inflammatory pathology of the airways that can be fed by a cytokine storm and result in severe respiratory failure (10% cases) and death (5%). The pathophysiological molecular mechanisms are currently not clearly defined. It is hypothesized that the transmembrane glycoprotein type II CD26, known for the enzyme activity Dipeptilpeptidase 4 of the extracellular domain, may play a main role in this condition. It is in fact considerably expressed at the level of parenchyma and pulmonary interstitium and carries out both systemic and paracrine enzymatic activity, modulating the function of various proinflammatory cytokines, growth factors and vasoactive peptides in the deep respiratory tract. Of particular interest is the fact that Dipeptilpeptidase 4 has been identified as a cellular receptor for S glycoprotein of MERS-COV. In the case of the SARS-COV 2 virus, the main receptor is the Angiotensin-Converting Enzyme 2 protein, but a possible interaction with Dipeptilpeptidase 4 also cannot be excluded. The selective blockade of Dipeptilpeptidase 4 could therefore favorably modulate the pulmonary inflammatory response in the subject affected by COVID-19. This protein is also known for the enzymatic degradation function of the native glucagon-like peptide 1, one of the main regulators of insulin secretion. This is why it is a molecular target in the treatment of diabetes (drugs that selectively inhibit Dipeptilpeptidase 4 are marketed with an indication for the treatment of type 2 diabetes). It is believed that the use of a Dipeptilpeptidase 4 inhibitor in people with diabetes and hospitalized for Covid-19 may be safe and of particular interest for an evaluation of the effects on laboratory and instrumental indicators of inflammatory lung disease. Among the drugs that selectively block Dipeptilpeptidase 4, the one with the greatest affinity is Sitagliptin.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled open label intervention study. Patients hospitalized for COVID-19 and affected by type 2 diabetes mellitus will be included in the study and divided into two groups by randomization: sitagliptin add-on standard of care therapy with nutritional therapy with or without insulin treatment (study group) vs nutritional therapy with or without insulin treatment (group of control, standard therapy). The design of the study provides an open randomization to allow its feasibility in times compatible with the achievement of adequate cases during the epidemic. The presence of placebo and a double-blind study, would lead to longer planning and enrollment times.

Patients with type 2 diabetes mellitus hospitalized for COVID-19 and randomized to the study group will be treated with sitagliptin at an adjusted dosage for estimated glomerular filtrate: 100 mg once daily (estimated glomerular filtration rate less than or equal to 45 mL / min / 1.73 m2) or 50 mg (estimated glomerular filtration rate 30-45 mL / min / 1.73 m2) in combination or not with insulin treatment. Patients with stage IV and V renal impairment (estimated glomerular filtration rate less than or equal to 30 mL / min / 1.73 m2) will be excluded. Enrolled patients will be followed according to the following scheme:

Time points:

* T0: The doctor explains the protocol to the patient and he gives to him the informed consent and the letter to the general practitioner.
* T1: The patient gives the signed and dated consent and officially enters the study. Basic assessments will be made. At the baseline, the clinical response, the main laboratory and instrumental tests will be taken into consideration. Biological samples will be taken for immunological study. Diabetic patients will begin treatment with Sitagliptin 100 or 50 mg add-on to nutritional therapy and, eventually, insulin treatment. Any other hypoglycemic agents taken before admission will be suspended.
* T2: 7 days after T1, for both groups of patients, evaluation of the clinical response, of the average daily blood glucose levels, of the main laboratory and instrumental tests.
* T3: 10 days after T2, for both groups of patients, evaluation of clinical response, average daily blood glucose levels, of the main laboratory and instrumental tests. Collection of biological samples for immunological study. End of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes, according to ADA 2020 criteria
* HbA1c levels at the entrance or in the two previous months <9%
* Diagnosis of Covid-19 (swab for positive SARS-COV2 RNA) with pneumonia, with or without increase in inflammation indexes, with or without respiratory failure
* No indication for tocilizumab therapy (BCRSS, Brescia Covid Respiratory Severity Scale, <3).
* Written and dated informed consent from the patient or his legally valid representative

Exclusion Criteria:

* Pregnancy
* Type 1 diabetes
* Stage IV and V renal failure (stimated glomerular filtration rate <30 ml / min)
* Treatment with Dipeptidyl peptidase-4 inhibitors or GLP-1 Receptor Agonists in the month prior to hospitalization
* Pioglitazone treatment in the month prior to hospitalization
* Treatment in the month preceding or in the course of hospitalization with "biological" drugs for immuno-rheumatological diseases (in particular tocilizumab)
* Presence of other acute or chronic ongoing infections
* Neurological or psychiatric diseases, diagnosis of hemoglobinopathy, diagnosis of liver disease, cancer, cystic fibrosis or malabsorption syndrome
* Dysphagia with need for artificial nutrition
* Positive history of acute and chronic pancreatitis
* Unstable cardiovascular disease or known atherosclerotic disease
* A history of alcohol or drug abuse
* Known human immunodeficiency virus (HIV) or hepatitis
* Presence of serious diseases or conditions that make the patient unsuitable for the study
* Surgery in the previous two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-12-29 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Time for clinical improvement | 1 month
  Evaluation of the time between randomization and two-point improvement on a seven-category scale (1, not hospitalized, return to normal activities; 2, not hospitalized, but unable to return to normal activities; 3, hospitalized without the need for oxygen therapy; 4, hospitalized, need for oxygen therapy; 5, hospitalized, need for non-invasive ventilatory support; 6, hospitalized, need for invasive mechanical ventilation or Extra Corporeal Membrane Oxygenation; 7, death)
Clinical parameter of acute lung disease | 1 month
  Clinical evaluation of the physiological parameter "cough" associated with acute lung disease from the start of the study to the end of the study.
Biochemical parameter of acute lung disease | 1 month
  Variation of biochemical parameter "glycemia" of acute lung disease from the beginning of the study to the end of study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "oxygen saturation by the use of a pulse oximeter" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "body temperature" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "respiratory rate" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "need for ventilatory support" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameters of acute lung disease | 1 month
  Variation of the clinical parameters "duration in days of ventilatory support, duration in days of oxygen therapy, duration in days of hospitalization, duration in days in the Intensive Care Unit, total length of stay in hospital" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "blood gas analysis" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "chest X ray" of acute lung disease from the beginning of the study to the end of the study.
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "PaO2/FiO2 ratio" of acute lung disease from the beginning of the study to the end of the study.
Biochemical parameter of acute lung disease | 1 month
  Variation of biochemical parameter "reactive C protein" of acute lung disease from the beginning of the study to the end of study.
Biochemical parameter of acute lung disease | 1 month
  Variation of biochemical parameter "blood count with formula" of acute lung disease from the beginning of the study to the end of study.
Biochemical parameter of acute lung disease | 1 month
  Variation of biochemical parameter "erythrocyte sedimentation rate" of acute lung disease from the beginning of the study to the end of study.
Biochemical parameter of acute lung disease | 1 month
  Variation of biochemical parameter "blood gas analysis" of acute lung disease from the beginning of the study to the end of study.
Biochemical parameter of acute lung disease | 1 month
  Variation of biochemical parameter "LDH" of acute lung disease from the beginning of the study to the end of study.

SECONDARY OUTCOMES:
Dipeptilpeptidase 4 expression in biological samples | 6 months
  The alteration of Dipeptilpeptidase 4 expression will be evaluated in the collected biological samples
Cytokine-inflammatory profile | 6 months
  Evaluation of inflammatory cytokines IL-2 and IL-7 in biological samples of treated patients and control group patients during infection.
Glycemic variability | 1 month
  Effect on glycemic variability by evaluating HbA1c levels.
Glycemic variability | 1 month
  Effect on glycemic variability by evaluating the average daily blood glucose levels.
Cytokine-inflammatory profile | 6 months
  Evaluation of the inflammatory cytokine granulocyte-colony stimulating factor in biological samples of treated patients and control group patients during infection.
Cytokine-inflammatory profile | 6 months
  Evaluation of the inflammatory cytokine interferon-γ inducible protein 10 in biological samples of treated patients and control group patients during infection.
Cytokine-inflammatory profile | 6 months
  Evaluation of the inflammatory cytokine monocyte chemoattractant protein 1 in biological samples of treated patients and control group patients during infection.
Cytokine-inflammatory profile | 6 months
  Evaluation of the inflammatory cytokine macrophage inflammatory protein 1-α in biological samples of treated patients and control group patients during infection.
Cytokine-inflammatory profile | 6 months
  Evaluation of the inflammatory cytokine tumour necrosis factor-α in biological samples of treated patients and control group patients during infection.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, PhD, Principal Investigator — University of Milan
Locations (1):
- ASST FBF Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang JK, Feng Y, Yuan MY, Yuan SY, Fu HJ, Wu BY, Sun GZ, Yang GR, Zhang XL, Wang L, Xu X, Xu XP, Chan JC. Plasma glucose levels and diabetes are independent predictors for mortality and morbidity in patients with SARS. Diabet Med. 2006 Jun;23(6):623-8. doi: 10.1111/j.1464-5491.2006.01861.x. PMID 16759303
- [Background] Perlman S, Azhar EI, Memish ZA, Hui DS, Zumla A. Confronting the persisting threat of the Middle East respiratory syndrome to global health security. Lancet Infect Dis. 2020 Feb;20(2):158-160. doi: 10.1016/S1473-3099(19)30347-0. Epub 2019 Jul 3. No abstract available. PMID 31279728
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Zou H, Zhu N, Li S. The emerging role of dipeptidyl-peptidase-4 as a therapeutic target in lung disease. Expert Opin Ther Targets. 2020 Feb;24(2):147-153. doi: 10.1080/14728222.2020.1721468. Epub 2020 Jan 31. PMID 31971463
- [Background] Meyerholz DK, Lambertz AM, McCray PB Jr. Dipeptidyl Peptidase 4 Distribution in the Human Respiratory Tract: Implications for the Middle East Respiratory Syndrome. Am J Pathol. 2016 Jan;186(1):78-86. doi: 10.1016/j.ajpath.2015.09.014. Epub 2015 Nov 18. PMID 26597880
- [Background] Ikeda T, Kumagai E, Iwata S, Yamakawa A. Soluble CD26/Dipeptidyl Peptidase IV Enhances the Transcription of IL-6 and TNF-alpha in THP-1 Cells and Monocytes. PLoS One. 2013 Jun 21;8(6):e66520. doi: 10.1371/journal.pone.0066520. Print 2013. PMID 23805228
- [Background] Raj VS, Mou H, Smits SL, Dekkers DH, Muller MA, Dijkman R, Muth D, Demmers JA, Zaki A, Fouchier RA, Thiel V, Drosten C, Rottier PJ, Osterhaus AD, Bosch BJ, Haagmans BL. Dipeptidyl peptidase 4 is a functional receptor for the emerging human coronavirus-EMC. Nature. 2013 Mar 14;495(7440):251-4. doi: 10.1038/nature12005. PMID 23486063
- [Background] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Background] Vankadari N, Wilce JA. Emerging WuHan (COVID-19) coronavirus: glycan shield and structure prediction of spike glycoprotein and its interaction with human CD26. Emerg Microbes Infect. 2020 Mar 17;9(1):601-604. doi: 10.1080/22221751.2020.1739565. eCollection 2020. PMID 32178593
- [Background] Kulcsar KA, Coleman CM, Beck SE, Frieman MB. Comorbid diabetes results in immune dysregulation and enhanced disease severity following MERS-CoV infection. JCI Insight. 2019 Oct 17;4(20):e131774. doi: 10.1172/jci.insight.131774. PMID 31550243
- [Background] Li K, Wohlford-Lenane CL, Channappanavar R, Park JE, Earnest JT, Bair TB, Bates AM, Brogden KA, Flaherty HA, Gallagher T, Meyerholz DK, Perlman S, McCray PB Jr. Mouse-adapted MERS coronavirus causes lethal lung disease in human DPP4 knockin mice. Proc Natl Acad Sci U S A. 2017 Apr 11;114(15):E3119-E3128. doi: 10.1073/pnas.1619109114. Epub 2017 Mar 27. PMID 28348219